CLINICAL TRIAL: NCT03292627
Title: Applying Non-invasive Hemodynamic Monitor to Predict the Risk of Perioperative Hypotension in Geriatric Patients Underwent Endoscopic Invasive Procedure
Brief Title: Non-invasive Monitor in Endoscopic Invasive Procedure
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201612030RINA
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2018-09

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde; Endoscopic Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mid age: mid age: 50-70 years old
  Interventions: Device: Portable Noninvasive Hemodynamic Monitor
- old age: old age: age older than 70 years old
  Interventions: Device: Portable Noninvasive Hemodynamic Monitor

INTERVENTIONS:
Device: Portable Noninvasive Hemodynamic Monitor — A non-invasive monitor for estimating patient's heart contractility and cardiac output by the change of thoracic electrical bioimpedance.
  Other Names: The ICON™ monitor

SUMMARY:
Investigators include the patients who need painless invasive endoscopic procedure, investigators collect the demographic data and apply the non-invasive device ICON on participants during the who procedure.

DETAILED DESCRIPTION:
Invasive endoscopy procedure including Endoscopic Retrograde Cholangio-Pancreatography (ERCP), endoscopic ultrasound guided fine needle aspiration (EUS-FNA), Endoscopic Retrograde Biliary Drainage (ERBD) and others is more and more popular which become the standard treatment before surgical intervention. However; the elder group who need this procedure is getting more common. The painless endoscopic sedation for elder group who has more comorbidity is not easy. During the procedure, the investigators found that the anticholinergic medication-buscopam which in order to suppress intestine mobilization can cause obvious tachycardia. Tachycardia makes the stroke volume decrease which enhance the perioperative hypotension, and the vasodilation effect of the analgesics make it worse.

Investigators are trying to find the non-invasive predictor of perioperative hypotension in geriatric group. Investigators collected the patients who need painless endoscopic invasive procedure, investigators will record their hemodynamic data including estimated cardiac output (CCO)，index of contractility (ICON)，NBP，HR，and saturation. Investigators also add the evaluation of frailty to evaluate the relationship between frailty and perioperative complications.

ELIGIBILITY:
Inclusion Criteria:

* patient who need painless endoscopic invasive procedures
* age above 50 y/o

Exclusion Criteria:

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators are trying to find the non-invasive predictor of perioperative hypotension in geriatric group. Investigator collected the patients who need painless endoscopic invasive procedure, investigator record their hemodynamic data including estimated cardiac output (CCO)，index of contractility (ICON)，NBP，HR，and saturation. Investigator wants to find that weather geriatric group has more risk of perioperative hypotension.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
ICON decrease 40% | during the painless procedure
  estimated index of contractility decrease 40%

SECONDARY OUTCOMES:
perioperative hypotension 40% | during the painless procedure
  BP decrease 40%

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-po Wang, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan